CLINICAL TRIAL: NCT05010759
Title: Stage 2B of: A Pivotal, Prospective, Three-Stage, Single-Arm Study of Focal Ablation of the Prostate With NanoTherm® Therapy System for a Limited-Volume, Clinically Localized, Intermediate-Risk Prostate Cancer
Brief Title: Study of Focal Ablation of the Prostate With NanoTherm® Therapy System for Intermediate-Risk Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment and company changing direction
Sponsor: MagForce USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGF-0115 - Stage 2B
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Ablation Arm (Experimental): Subjects in this arm of the study will have focal ablation of the prostate cancer lesion with the NanoTherm technology. This ablation will be followed-up transperineal prostate biopsy at 4 months after treatment.
  Interventions: Device: NanoTherm Ablation

INTERVENTIONS:
Device: NanoTherm Ablation — Iron nanoparticles are instilled into the prostate cancer lesion and then the particles are heated using a magnetic field and this heating ablates the prostate cancer lesion.

SUMMARY:
Stage 2B: NanoTherm ablation of focal prostate cancer in small lesions in Gleason 3+4 disease. The outcome of this ablation is validated by a transperineal biopsy at 4 months after ablation.

DETAILED DESCRIPTION:
Presently, patients having intermediate-risk prostate carcinoma have to make a very difficult decision regarding treatment, as active surveillance will not immediately alter the current quality of life. However, because there is a risk of progressive disease or due to patient anxiety due to an untreated tumor, many patients opt for active treatment, often using radiation or prostatectomy, and sometimes in combination with androgen deprivation. Unfortunately, radiation, surgery, and androgen deprivation have multiple and potentially profound side effects including sexual, urinary, and bowel complications. As a small fraction of men dies from this disease, the number of men needed to treat to prevent one death is large, resulting in many men with side effects or complications to help prevent the one death. It is for these reasons that there is a major need for focal therapy for this group of patients who most commonly are treated actively with surgery or radiation; such focal therapy could ablate the detected tumor(s) within the prostate, control the disease while avoiding side effects of whole gland therapies and controlling tumor growth within the prostate detected by (multiparameter-) MRI and histopathologically confirmed by biopsy. MagForce NanoTherm® Therapy offers this option by noninvasive ablation of small tumors in a 1-2 ml target volume of the prostate, a treatment that is not possible with any other technology on the market.

This study evaluates the use of NanoTherm ablation as a method of treating these intermediate grade lesions allowing patients to return to active surveillance without definitive treatment such as external beam radiation or prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 85
* Male
* Prostate adenocarcinoma on biopsy
* Clinical stage T1c/T2a/T2b, N0, M0/Mx with no lesion larger than 2cc in volume
* The following biopsy findings (biopsy must have MRI visualization and be within 6 months of planned NanoTherm® treatment):

  * A positive biopsy for prostate cancer from the MRI-visualized lesion, at least one of which must be Gleason 3+4 (grade group 2)
* Lesion must be visualized by Multiparametric Magnetic Resonance Imaging (MP-MRI) on a scan that is less than 6 months old
* Patient expresses a preference for active surveillance, rather than surgery or radiation, to manage prostate cancer
* Based on the evaluation of the study investigator, appropriate for instillation of NanoTherm® under anesthesia based on location and size of the clinical target volume (CTV)

Exclusion Criteria:

* Previous treatment for cancer with radiation, androgen deprivation (including LHRH-agonists or antagonists or antiandrogens), or surgery for prostate cancer
* Active urinary tract infection
* Metallic implants below the neck
* Gleason 3+4 or higher cancer on prostate biopsy outside of the planned CTV
* Gleason 4+3 or higher on any prostate biopsy
* Hematological abnormality indicating increased risk of bleeding or clotting, for example low platelet count or anemia
* Participation concurrently in another clinical trial for prostate disease or in the last 30 days
* Known hypersensitivity to Axumin®

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Rate of Ablation Success | 4 months (+/- 1 Month)
  Rate of subjects with a biopsy confirmed ablation of prostate cancer lesion

SECONDARY OUTCOMES:
Adverse Event Rate | 4 months (+/- 1 Month)
  Rate of Adverse Events of Special Interest (AESI)

CONTACTS AND LOCATIONS:
Overall Officials: David Hammond, MS, Study Director — MagForce USA
Locations (4):
- United States (4):
  - Florida Urology Partners, Tampa, Florida
  - Urology Austin, Austin, Texas
  - MagForce - San Antonio, San Antonio, Texas
  - MagForce USA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No